CLINICAL TRIAL: NCT00600106
Title: WISE Ancillary Study Data Analyses: Efficacy of Hormone Replacement on Myocardial Ischemia in Postmenopausal Women With Normal/Minimal Coronary Artery Disease: Data Analysis
Brief Title: Data Analyses for Ancillary WISE Femhrt Hormone Replacement Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Parke-Davis (Industry); University of Pittsburgh (Other); University of Florida (Other); Allegheny University (Unknown); University of Alabama at Birmingham (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9260; IRB#0505140 (Other: University of Pittsburgh)
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hormone replacement therapy (Active Comparator): Hormone replacement therapy with 1 mg norethindrone/10 mcg thinyl estradiol (1/10 NA/EE)
  Interventions: Drug: 1/10 NA/EE
- Placebo (Placebo Comparator): 1mg placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1/10 NA/EE — Hormone replacement therapy with 1 mg norethindrone/10 mcg thinyl estradiol (1/10 NA/EE)
  Arms: Hormone replacement therapy
Drug: Placebo — 1 mg placebo
  Arms: Placebo

SUMMARY:
The goal of the main trial was to evaluate the effect of low dose hormone replacement therapy with 1 mg norethindrone/10mcg ethinyl estradiol in postmenopausal women with a history of chest discomfort, myocardial ischemia and no obstructive CAD. For the purposes of this study as a core lab coordinating center, the investigators will be performing P31 MRS core lab analyses; hormone core lab analyses; lipid core lab analyses; glucose, insulin and HOMA core lab analyses; exercise stress test/Holter monitor core lab analyses; brachial artery reactivity test core lab analyses; full study data analyses for manuscript preparation and the writing and submission and publication of manuscript.

The main trial duration: December 1999 - May 2003.

The ancillary data analysis project duration: April 2006 - March 2010.

DETAILED DESCRIPTION:
See Brief Summary above.

ELIGIBILITY:
Inclusion Criteria

* Postmenopausal WISE and nonWISE study participants
* Normal/minimally diseased coronary arteries (<50% luminal diameter stenosis in all epicardial coronary arteries) within 36 months of ancillary study entry and no intercurrent MI, PTCA, CABG
* Any one (or multiple) of the following criteria suggestive of myocardial ischemia within 36 months of ancillary study entry:

  1. Abnormal P-31 magnetic resonance spectroscopy (a fall in quantitative PCr/ATP ratio >15% from control) performed at a WISE or nonWISE site
  2. Positive exercise stress test (> or = 1mm horizontal or downsloping, or > or =1.5mm upsloping ST segment depression measured 0.08 msec after the J point), performed and/or interpretated by a WISE or WISE ancillary ancillary trial investigator
  3. Reversible stress radionuclide perfusion defect > equivocal and not attributable to breast/imaging artifact. performed as part of the WISE protocol
  4. Coronary artery flow reserve <2.25 performed. as part of using the WISE protocol
* No contraindications to 12 weeks of FemHRT or hormone replacement therapy
* Normal mammogram and pelvic exam (including PAP smear for those with an intact uterus) within 12 months of study entry
* Documented normal liver function testing (SGOT) within 3 months of study entry.

Exclusion Criteria

* Documented myocardial infarction, coronary artery bypass surgery or mechanical revascularization
* Systolic blood pressure >200 mmHg or diastolic blood pressure >105 mmHg
* LDL-cholesterol >190 mg/dl, triglycerides > or = 300 mg/dl
* Clinically significant hepatic or renal dysfunction (SGOT more than 1.2 times normal at baseline, serum creatinine >2)
* Uncontrolled diabetes mellitus (FBS > or = 225 mg/dl) or new onset diabetes until stabilized
* Clinically significant valvular heart disease, dilated cardiomyopathy, or congestive heart failure (NYHA Class IV or severe Class III)
* Currently on hormone replacement therapy and unwilling/unable to withdraw treatment prior to study, (participants are eligible for study entry 4-8 weeks following hormone replacement therapy withdrawal, at the discretion of the WISE ancillary trial Principal Investigator)
* Previous breast cancer, mammogram suggestive of cancer, or endometrial cancer without hysterectomy
* Abnormal uterine bleeding or abnormal Pap smear (SIL I, II or III, carcinoma in situ, or cancer)
* Previous deep venous thrombosis, pulmonary embolism, or other thromboembolic disorder.
* Alcoholism or drug abuse
* Participation in any other investigational drug or device study

Women with elevated diastolic (> or = 90 mm Hg) or systolic (> or = 140 mm Hg) blood pressure, LDL-cholesterol (> or = 160 mg/dl), fasting blood sugar (> or = 130 mg/dl) and women who smoke cigarettes will be told their risk factor levels and referred for evaluation and treatment by their private physician.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 1999-12; Primary Completion 2003-05 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Noel Bairey Merz, MD, Study Chair — Cedars-Sinai Medical Center; Carl Pepine, MD, Principal Investigator — University of Florida; Steve Reis, MD, Principal Investigator — University of Pittsburgh; Nathaniel Reichek, MD, Principal Investigator — Allegheny University of the Health Sciences; William Rogers, MD, Principal Investigator — University of Alabama at Birmingham; Vijay Misra, MD, Principal Investigator — University of Alabama at Birmingham; Robert B Weiss, MD, Principal Investigator — Johns Hopkins University; Sheryl Kelsey, PhD, Principal Investigator — University of Pittsburgh; George Sopko, MD, Study Director — National Institute of Health (WISE Project Officer); James Symons, PhD, Study Director — Parke-Davis; Connie McLaughlin, PharmD, Study Director — Parke-Davis
Locations (1):
- Cedars-Sinai Women's Heart Center, 8631 W. 3rd St, Suite 740, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panza JA. Myocardial ischemia and the pains of the heart. N Engl J Med. 2002 Jun 20;346(25):1934-5. doi: 10.1056/NEJMp020047. No abstract available. PMID 12075053
- [Background] Cannon RO 3rd. Does coronary endothelial dysfunction cause myocardial ischemia in the absence of obstructive coronary artery disease? Circulation. 1997 Nov 18;96(10):3251-4. No abstract available. PMID 9396408
- [Background] Williams JK, Adams MR, Klopfenstein HS. Estrogen modulates responses of atherosclerotic coronary arteries. Circulation. 1990 May;81(5):1680-7. doi: 10.1161/01.cir.81.5.1680. PMID 2331772
- [Background] Williams JK, Shively CA, Clarkson TB. Determinants of coronary artery reactivity in premenopausal female cynomolgus monkeys with diet-induced atherosclerosis. Circulation. 1994 Aug;90(2):983-7. doi: 10.1161/01.cir.90.2.983. PMID 8044971
- [Background] Gilligan DM, Quyyumi AA, Cannon RO 3rd. Effects of physiological levels of estrogen on coronary vasomotor function in postmenopausal women. Circulation. 1994 Jun;89(6):2545-51. doi: 10.1161/01.cir.89.6.2545. PMID 8205663
- [Background] Reis SE, Gloth ST, Blumenthal RS, Resar JR, Zacur HA, Gerstenblith G, Brinker JA. Ethinyl estradiol acutely attenuates abnormal coronary vasomotor responses to acetylcholine in postmenopausal women. Circulation. 1994 Jan;89(1):52-60. doi: 10.1161/01.cir.89.1.52. PMID 8281693
- [Background] Merz CN, Kelsey SF, Pepine CJ, Reichek N, Reis SE, Rogers WJ, Sharaf BL, Sopko G. The Women's Ischemia Syndrome Evaluation (WISE) study: protocol design, methodology and feasibility report. J Am Coll Cardiol. 1999 May;33(6):1453-61. doi: 10.1016/s0735-1097(99)00082-0. PMID 10334408
- [Background] Sharaf BL, Pepine CJ, Kerensky RA, Reis SE, Reichek N, Rogers WJ, Sopko G, Kelsey SF, Holubkov R, Olson M, Miele NJ, Williams DO, Merz CN; WISE Study Group. Detailed angiographic analysis of women with suspected ischemic chest pain (pilot phase data from the NHLBI-sponsored Women's Ischemia Syndrome Evaluation [WISE] Study Angiographic Core Laboratory). Am J Cardiol. 2001 Apr 15;87(8):937-41; A3. doi: 10.1016/s0002-9149(01)01424-2. PMID 11305981
- [Background] The manual of laboratory operations 1. Lipid and lipoprotein analysis. Bethesda: Lipid Research Clinics Program. National Institutes of Health. DHEW Publication No. 75-628; 1974.
- [Background] Barrett-Connor E, Goodman-Gruen D. Prospective study of endogenous sex hormones and fatal cardiovascular disease in postmenopausal women. BMJ. 1995 Nov 4;311(7014):1193-6. doi: 10.1136/bmj.311.7014.1193. PMID 7488894
- [Background] Helmer DC, Ragland DR, Syme SL. Hostility and coronary artery disease. Am J Epidemiol. 1991 Jan 15;133(2):112-22. doi: 10.1093/oxfordjournals.aje.a115850. PMID 1985442
- [Background] Naughton MJ, Shumaker SA, Anderson RT, et al. Psychological aspects of health-related quality of life measurement: tests and scales. Philadelphia: Lippincott-Raven Publishers; 1996.
- [Background] MANDLER G, MANDLER JM, UVILLER ET. Autonomic feedback: the perception of autonomic activity. J Abnorm Psychol. 1958 May;56(3):367-73. doi: 10.1037/h0048083. No abstract available. PMID 13538604
- [Background] Ware JE, Kosinski M, Gandek B. SF-36 Health Survey. Manual and interpretation guide. Lincoln: Quality Metric Inc.; 1993.
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Hilditch JR, Lewis J, Peter A, van Maris B, Ross A, Franssen E, Guyatt GH, Norton PG, Dunn E. A menopause-specific quality of life questionnaire: development and psychometric properties. Maturitas. 1996 Jul;24(3):161-75. doi: 10.1016/s0378-5122(96)82006-8. PMID 8844630
- [Background] Rosano GM, Sarrel PM, Poole-Wilson PA, Collins P. Beneficial effect of oestrogen on exercise-induced myocardial ischaemia in women with coronary artery disease. Lancet. 1993 Jul 17;342(8864):133-6. doi: 10.1016/0140-6736(93)91343-k. PMID 8101254
- [Background] Olson MB, Kelsey SF, Matthews K, Shaw LJ, Sharaf BL, Pohost GM, Cornell CE, McGorray SP, Vido D, Bairey Merz CN. Symptoms, myocardial ischaemia and quality of life in women: results from the NHLBI-sponsored WISE Study. Eur Heart J. 2003 Aug;24(16):1506-14. doi: 10.1016/s0195-668x(03)00279-3. PMID 12919775
- [Background] Albertsson PA, Emanuelsson H, Milsom I. Beneficial effect of treatment with transdermal estradiol-17-beta on exercise-induced angina and ST segment depression in syndrome X. Int J Cardiol. 1996 Apr 19;54(1):13-20. doi: 10.1016/0167-5273(96)02560-0. PMID 8792180
- [Background] Adamson DL, Webb CM, Collins P. Esterified estrogens combined with methyltestosterone improve emotional well-being in postmenopausal women with chest pain and normal coronary angiograms. Menopause. 2001 Jul-Aug;8(4):233-8. doi: 10.1097/00042192-200107000-00003. PMID 11449079
- [Background] Rosano GM, Peters NS, Lefroy D, Lindsay DC, Sarrel PM, Collins P, Poole-Wilson PA. 17-beta-Estradiol therapy lessens angina in postmenopausal women with syndrome X. J Am Coll Cardiol. 1996 Nov 15;28(6):1500-5. doi: 10.1016/s0735-1097(96)00348-8. PMID 8917264
- [Background] Gerhard M, Walsh BW, Tawakol A, Haley EA, Creager SJ, Seely EW, Ganz P, Creager MA. Estradiol therapy combined with progesterone and endothelium-dependent vasodilation in postmenopausal women. Circulation. 1998 Sep 22;98(12):1158-63. doi: 10.1161/01.cir.98.12.1158. PMID 9743505
- [Background] Herrington DM, Werbel BL, Riley WA, Pusser BE, Morgan TM. Individual and combined effects of estrogen/progestin therapy and lovastatin on lipids and flow-mediated vasodilation in postmenopausal women with coronary artery disease. J Am Coll Cardiol. 1999 Jun;33(7):2030-7. doi: 10.1016/s0735-1097(99)00128-x. PMID 10362210
- [Background] Koh KK, Cardillo C, Bui MN, Hathaway L, Csako G, Waclawiw MA, Panza JA, Cannon RO 3rd. Vascular effects of estrogen and cholesterol-lowering therapies in hypercholesterolemic postmenopausal women. Circulation. 1999 Jan 26;99(3):354-60. doi: 10.1161/01.cir.99.3.354. PMID 9918521
- [Background] Herrington DM, Reboussin DM, Brosnihan KB, Sharp PC, Shumaker SA, Snyder TE, Furberg CD, Kowalchuk GJ, Stuckey TD, Rogers WJ, Givens DH, Waters D. Effects of estrogen replacement on the progression of coronary-artery atherosclerosis. N Engl J Med. 2000 Aug 24;343(8):522-9. doi: 10.1056/NEJM200008243430801. PMID 10954759
- [Background] Hulley S, Grady D, Bush T, Furberg C, Herrington D, Riggs B, Vittinghoff E. Randomized trial of estrogen plus progestin for secondary prevention of coronary heart disease in postmenopausal women. Heart and Estrogen/progestin Replacement Study (HERS) Research Group. JAMA. 1998 Aug 19;280(7):605-13. doi: 10.1001/jama.280.7.605. PMID 9718051
- [Background] Waters DD, Alderman EL, Hsia J, Howard BV, Cobb FR, Rogers WJ, Ouyang P, Thompson P, Tardif JC, Higginson L, Bittner V, Steffes M, Gordon DJ, Proschan M, Younes N, Verter JI. Effects of hormone replacement therapy and antioxidant vitamin supplements on coronary atherosclerosis in postmenopausal women: a randomized controlled trial. JAMA. 2002 Nov 20;288(19):2432-40. doi: 10.1001/jama.288.19.2432. PMID 12435256
- [Background] Lobo RA. Evaluation of cardiovascular event rates with hormone therapy in healthy, early postmenopausal women: results from 2 large clinical trials. Arch Intern Med. 2004 Mar 8;164(5):482-4. doi: 10.1001/archinte.164.5.482. No abstract available. PMID 15006823
- [Background] Rossouw JE, Prentice RL, Manson JE, Wu L, Barad D, Barnabei VM, Ko M, LaCroix AZ, Margolis KL, Stefanick ML. Postmenopausal hormone therapy and risk of cardiovascular disease by age and years since menopause. JAMA. 2007 Apr 4;297(13):1465-77. doi: 10.1001/jama.297.13.1465. PMID 17405972
- [Background] Campisi R, Nathan L, Pampaloni MH, Schoder H, Sayre JW, Chaudhuri G, Schelbert HR. Noninvasive assessment of coronary microcirculatory function in postmenopausal women and effects of short-term and long-term estrogen administration. Circulation. 2002 Jan 29;105(4):425-30. doi: 10.1161/hc0402.102860. PMID 11815423
- [Background] Johnson BD, Shaw LJ, Buchthal SD, Bairey Merz CN, Kim HW, Scott KN, Doyle M, Olson MB, Pepine CJ, den Hollander J, Sharaf B, Rogers WJ, Mankad S, Forder JR, Kelsey SF, Pohost GM; National Institutes of Health-National Heart, Lung, and Blood Institute. Prognosis in women with myocardial ischemia in the absence of obstructive coronary disease: results from the National Institutes of Health-National Heart, Lung, and Blood Institute-Sponsored Women's Ischemia Syndrome Evaluation (WISE). Circulation. 2004 Jun 22;109(24):2993-9. doi: 10.1161/01.CIR.0000130642.79868.B2. Epub 2004 Jun 14. PMID 15197152
- [Background] Buchthal SD, den Hollander JA, Merz CN, Rogers WJ, Pepine CJ, Reichek N, Sharaf BL, Reis S, Kelsey SF, Pohost GM. Abnormal myocardial phosphorus-31 nuclear magnetic resonance spectroscopy in women with chest pain but normal coronary angiograms. N Engl J Med. 2000 Mar 23;342(12):829-35. doi: 10.1056/NEJM200003233421201. PMID 10727587
- [Background] Halcox JP, Schenke WH, Zalos G, Mincemoyer R, Prasad A, Waclawiw MA, Nour KR, Quyyumi AA. Prognostic value of coronary vascular endothelial dysfunction. Circulation. 2002 Aug 6;106(6):653-8. doi: 10.1161/01.cir.0000025404.78001.d8. PMID 12163423
- [Background] Kaski JC, Rosano GM, Collins P, Nihoyannopoulos P, Maseri A, Poole-Wilson PA. Cardiac syndrome X: clinical characteristics and left ventricular function. Long-term follow-up study. J Am Coll Cardiol. 1995 Mar 15;25(4):807-14. doi: 10.1016/0735-1097(94)00507-M. PMID 7884081
- [Background] Kemp HG, Kronmal RA, Vlietstra RE, Frye RL. Seven year survival of patients with normal or near normal coronary arteriograms: a CASS registry study. J Am Coll Cardiol. 1986 Mar;7(3):479-83. doi: 10.1016/s0735-1097(86)80456-9. PMID 3512658
- [Background] Lichtlen PR, Bargheer K, Wenzlaff P. Long-term prognosis of patients with anginalike chest pain and normal coronary angiographic findings. J Am Coll Cardiol. 1995 Apr;25(5):1013-8. doi: 10.1016/0735-1097(94)00519-v. PMID 7897110
- [Background] Shaw LJ, Merz CN, Pepine CJ, Reis SE, Bittner V, Kip KE, Kelsey SF, Olson M, Johnson BD, Mankad S, Sharaf BL, Rogers WJ, Pohost GM, Sopko G; Women's Ischemia Syndrome Evaluation (WISE) Investigators. The economic burden of angina in women with suspected ischemic heart disease: results from the National Institutes of Health--National Heart, Lung, and Blood Institute--sponsored Women's Ischemia Syndrome Evaluation. Circulation. 2006 Aug 29;114(9):894-904. doi: 10.1161/CIRCULATIONAHA.105.609990. Epub 2006 Aug 21. PMID 16923752
- [Background] Johnson BD, Shaw LJ, Pepine CJ, Reis SE, Kelsey SF, Sopko G, Rogers WJ, Mankad S, Sharaf BL, Bittner V, Bairey Merz CN. Persistent chest pain predicts cardiovascular events in women without obstructive coronary artery disease: results from the NIH-NHLBI-sponsored Women's Ischaemia Syndrome Evaluation (WISE) study. Eur Heart J. 2006 Jun;27(12):1408-15. doi: 10.1093/eurheartj/ehl040. Epub 2006 May 23. PMID 16720691
- [Background] von Mering GO, Arant CB, Wessel TR, McGorray SP, Bairey Merz CN, Sharaf BL, Smith KM, Olson MB, Johnson BD, Sopko G, Handberg E, Pepine CJ, Kerensky RA; National Heart, Lung, and Blood Institute. Abnormal coronary vasomotion as a prognostic indicator of cardiovascular events in women: results from the National Heart, Lung, and Blood Institute-Sponsored Women's Ischemia Syndrome Evaluation (WISE). Circulation. 2004 Feb 17;109(6):722-5. doi: 10.1161/01.CIR.0000115525.92645.16. PMID 14970106
- [Background] Lanza GA, Colonna G, Pasceri V, Maseri A. Atenolol versus amlodipine versus isosorbide-5-mononitrate on anginal symptoms in syndrome X. Am J Cardiol. 1999 Oct 1;84(7):854-6, A8. doi: 10.1016/s0002-9149(99)00450-6. PMID 10513787
- [Background] Lerman A, Burnett JC Jr, Higano ST, McKinley LJ, Holmes DR Jr. Long-term L-arginine supplementation improves small-vessel coronary endothelial function in humans. Circulation. 1998 Jun 2;97(21):2123-8. doi: 10.1161/01.cir.97.21.2123. PMID 9626172
- [Background] Cannon RO 3rd, Quyyumi AA, Mincemoyer R, Stine AM, Gracely RH, Smith WB, Geraci MF, Black BC, Uhde TW, Waclawiw MA, et al. Imipramine in patients with chest pain despite normal coronary angiograms. N Engl J Med. 1994 May 19;330(20):1411-7. doi: 10.1056/NEJM199405193302003. PMID 8159194
- [Background] Eriksson BE, Tyni-Lenne R, Svedenhag J, Hallin R, Jensen-Urstad K, Jensen-Urstad M, Bergman K, Selven C. Physical training in Syndrome X: physical training counteracts deconditioning and pain in Syndrome X. J Am Coll Cardiol. 2000 Nov 1;36(5):1619-25. doi: 10.1016/s0735-1097(00)00931-1. PMID 11079667
- [Result] Rossouw JE, Anderson GL, Prentice RL, LaCroix AZ, Kooperberg C, Stefanick ML, Jackson RD, Beresford SA, Howard BV, Johnson KC, Kotchen JM, Ockene J; Writing Group for the Women's Health Initiative Investigators. Risks and benefits of estrogen plus progestin in healthy postmenopausal women: principal results From the Women's Health Initiative randomized controlled trial. JAMA. 2002 Jul 17;288(3):321-33. doi: 10.1001/jama.288.3.321. PMID 12117397
- [Derived] Merz CN, Olson MB, McClure C, Yang YC, Symons J, Sopko G, Kelsey SF, Handberg E, Johnson BD, Cooper-DeHoff RM, Sharaf B, Rogers WJ, Pepine CJ. A randomized controlled trial of low-dose hormone therapy on myocardial ischemia in postmenopausal women with no obstructive coronary artery disease: results from the National Institutes of Health/National Heart, Lung, and Blood Institute-sponsored Women's Ischemia Syndrome Evaluation (WISE). Am Heart J. 2010 Jun;159(6):987.e1-7. doi: 10.1016/j.ahj.2010.03.024. PMID 20569710

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hormone Replacement Therapy | Placebo
Started | 18 | 19
Completed | 17 | 18
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hormone Replacement Therapy | Placebo | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9) | 59 (7) | 57.5 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Nonwhite | 3 | 3 | 6
  White | 15 | 16 | 31
Education [Number; unit: participants]
  High school or less | 10 | 13 | 23
  College | 8 | 6 | 14
Current HT use prior to entry [Number; unit: participants]
  Current HT use prior to entry | 6 | 8 | 14
  No HT prior to entry | 12 | 11 | 23
History of Hypertension [Number; unit: participants]
  Hypertension | 5 | 14 | 19
  Normal blood pressure | 13 | 5 | 18
History of Diabetes [Number; unit: participants]
  History of Diabetes | 4 | 5 | 9
  No Diabetes | 14 | 14 | 28
History of Dyslipidemia [Number; unit: participants]
  Dyslipidemia | 11 | 7 | 18
  Normal values | 7 | 12 | 19
Current Smoking [Number; unit: participants]
  Smoking | 2 | 2 | 4
  No smoking | 16 | 17 | 33
Total Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 195 (47) | 205 (39) | 200 (43)
HDL-Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 48 (16) | 54 (9) | 51 (12.5)
LDL-Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 120 (51) | 124 (38) | 122 (44.5)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 132 (92) | 134 (64) | 133 (78)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 130 (18) | 136 (18) | 133 (18)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 76 (13) | 78 (9) | 77 (11)
Pulse [Mean (Standard Deviation); unit: beats per minute] | 68 (8) | 76 (11) | 72 (9.5)
Fasting Blood Sugar [Mean (Standard Deviation); unit: mg/dl] | 93 (17) | 94 (20) | 93.5 (18.5)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31 (9) | 31 (7) | 31 (8)
Waist circumference [Mean (Standard Deviation); unit: cm.] | 92 (17) | 93 (15) | 92.5 (16)

OUTCOME MEASURES:

1. Primary Outcome: Inducible Myocardial Ischemia
Description: Inducible myocardial ischemia measured by P-31 gated magnetic resonance cardiac spectroscopy (MRS) is reported as change (∆) in PCr/ATP ratio, with isometric submaximal handgrip stress. PCr/ATP ratio defined as (stress-[average of rest and recovery periods]) / average of rest and recover periods X 100, and expressed as % mean ± SD. For this trial, myocardial ischemia was pre-specified as a fall in quantitative PCR/ATP ratio >20% from rest, and a lower value is considered indicative of greater ischemia.
Time Frame: Baseline
Population: Among the 35 women, 28 baseline and 26 exit MRS results were technically adequate for spectral analyses with rest, handgrip exercise, and recovery spectra. A total of 24 women (13 drug, 11 placebo) had both baseline and exit P31's.
Measure: Mean (Standard Deviation); unit: percent changed in PCR/ATP ratio
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 15 | 13
percent changed in PCR/ATP ratio | -13.8 (24.2) | -7.0 (22.8)
Statistical Analysis 1: Comparison: Hormone Replacement Therapy vs Placebo; Data were presented in tables as means and SDs for continuous variables and frequencies for categorical variables. Comparisons between the placebo and 1/10 NA/EE groups were don using Wilcoxon rank sum test for continuous measurement and Fisher's exact test for discrete data. The strategy of analysis was "intention to treat" with comparing the study groups in term of treatment to which they were randomly allocated; Test type: Superiority or Other — All tests were two-sided with p values <0.05; p = 0.36, t-test (nonparametric Wilcoxon test)

2. Secondary Outcome: Physical Functional Disability - Functional Capacity (METs)
Description: Physical functional disability measured by exercise stress testing. Functional capacity was measured as metabolism equivalents (METs), exercise duration, and exercise-induced chest pain. A MET is defined as the resting metabolic rate, that is, the amount or oxygen consumet at rest, sitting quietly in a chair, approximately 3.5 ml O2 / kg / min (1.2 kcallmin for a 70-kg person). As such, work at METs requires twice the resting metabolism or 7.0 ml O2/kg/min, and so on.
Time Frame: Baseline
Population: Exercise stress testing at baseline by treatment
Measure: Mean (Standard Deviation); unit: metabolism equivalents
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 17 | 16
metabolism equivalents | 5.4 (2.6) | 5.4 (1.8)
Statistical Analysis 1: Comparison: Hormone Replacement Therapy vs Placebo; Test type: Superiority or Other; p = 0.93, Wilcoxon rank sum test

3. Primary Outcome: Endothelial Dysfunction (FMD)
Description: Endothelial dysfunction refers to altered vasoactive, anticoagulant, and anti-inflammatory properties of endothelium, and dysregulated vascular growth remodeling that results from a loss of nitric oxide (NO) bioactivity in the endothelium. Brachial Artery Reactivity Testing (BART), high-frequency ultrasonographic imaging of the brachial artery, evaluates flow-mediated vasodilation (FMD), an endothelium-dependent function. The technique provokes the release of nitric oxide, resulting in vasodilation that can be quantitated as an index of endothelial dysfunction.
  Flow-mediated vasodilation is typically expressed as the change in post-stimulus diameter as a percentage of the baseline diameter [diameter after cuff deflation - baseline diameter / baseline diameter) x 100].
Time Frame: Baseline
Population: Brachial artery reactivity testing at baseline by treatment
Measure: Mean (Standard Deviation); unit: percentage of pre-stimulus diameter
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 16 | 18
percentage of pre-stimulus diameter | 8.2 (7.8) | 8.8 (7.3)
Statistical Analysis 1: Comparison: Hormone Replacement Therapy vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other — All tests were two-sided with p values <0.05; p = 0.77, Wilcoxon rank sum test

4. Secondary Outcome: Quality of Life - Menopause Symptoms
Description: Quality of life assessed by menopausal symptoms and psychological questionnaires
Time Frame: Baseline
Population: Menopause Symptoms at baseline by treatment
Measure: Number; unit: percent of participants
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 18 | 19
percent of participants
  Hot flushes or flashing | 89 | 68
  Poor memory | 76 | 53
  Change in sexual desire | 50 | 37
  Vaginal dryness | 44 | 58
  Avoiding intimacy | 39 | 37

5. Primary Outcome: Endothelial Dysfunction (FMD)
Description: Endothelial dysfunction refers to altered vasoactive, anticoagulant, and anti-inflammatory properties of endothelium, and dysregulated vascular growth remodeling that results from a loss of nitric oxide (NO) bioactivity in the endothelium. Brachial Artery Reactivity Testing (BART), high-frequency ultrasonographic imaging of the brachial artery, evaluates flow-mediated vasodilation (FMD), an endothelium-dependent function. The technique provokes the release of nitric oxide, resulting in vasodilation that can be quantitated as an index of vasomotor function.
  Flow-mediated vasodilation is typically expressed as the change in post-stimulus diameter as a percentage of the baseline diameter [diameter after cuff deflation - baseline diameter / baseline diameter) x 100].
Time Frame: 12 weeks
Population: Brachial artery reactivity testing at study exit by treatment
Measure: Mean (Standard Deviation); unit: percentage of pre-stimulus diameter
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 15 | 16
percentage of pre-stimulus diameter | 8.8 (5.3) | 7.3 (6.1)
Statistical Analysis 1: Comparison: Hormone Replacement Therapy vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other — All tests were two-sided with p values <0.05; p = 0.38, Wilcoxon rank sum test

6. Secondary Outcome: Quality of Life - Menopause Symptoms
Description: Quality of life assessed by menopausal symptoms and psychological questionnaires
Time Frame: 12 weeks
Population: Menopause Symptoms at exit by treatment
Measure: Number; unit: percent of participants
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 17 | 18
percent of participants
  Hot flushes or flashing | 41 | 89
  Poor memory | 59 | 78
  Change in sexual desire | 35 | 67
  Vaginal dryness | 35 | 67
  Avoiding intimacy | 24 | 56

7. Secondary Outcome: Quality of Life - Health Survey
Description: Quality of life assessed by cardiac symptoms and psychological questionnaires (SF 36 scale - Short Form Health Survey) The SF-36 includes one multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions.
  Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Baseline
Population: SF-36 scale at baseline by treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 18 | 19
units on a scale
  Physical functioning | 60.8 (27.5) | 43.8 (27.4)
  Role-physical | 54.2 (41.3) | 37.3 (40.2)
  Role-emotional | 70.3 (42.6) | 66.7 (41.6)
  Bodily pain | 53.3 (21.4) | 42.1 (17.4)
  General health | 55.4 (19.4) | 57.4 (15.1)
  Mental health | 66.7 (20.6) | 65.7 (19.9)
  Vitality | 35.6 (23.1) | 42.9 (20.4)
  Social functioning | 59.4 (14.7) | 53.2 (24.3)

8. Secondary Outcome: Quality of Life - Health Survey
Description: as for outcome 7
Time Frame: 12 weeks
Population: SF-36 scale at exit by treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 17 | 18
units on a scale
  Physical functioning | 59.4 (23.5) | 44.4 (29.5)
  Role-physical | 58.8 (37.4) | 25.0 (33.2)
  Role-emotional | 76.5 (34.9) | 66.7 (39.6)
  Bodily pain | 54.5 (23.6) | 41.5 (21.6)
  General health | 55.2 (19.7) | 57.2 (15.8)
  Mental health | 66.4 (19.6) | 69.3 (18.8)
  Vitality | 35.6 (24.5) | 41.2 (18.0)
  Social functioning | 59.4 (16.0) | 56.1 (20.6)

9. Primary Outcome: Inducible Myocardial Ischemia
Description: as for outcome 1
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change in PCR/ATP ratio
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 14 | 12
percent change in PCR/ATP ratio | -7.7 (20.8) | 1.1 (9.7)
Statistical Analysis 1: Comparison: Hormone Replacement Therapy vs Placebo; Data were presented in tables as means and SDs for continuous variables and frequencies for categorical variables. Comparisons between the placebo and 1/10 NA/EE groups were don using Wilcoxon rank sum test for continuous measurement and Fisher's exact test for discrete data. The strategy of analysis was "intention to treat" with comparing the study groups in term of treatment to which they were randomly allocated. All tests were two-sided with p values <0.05; Test type: Superiority or Other; p = 0.17, t-test (nonparametric Wilcoxon test)

10. Secondary Outcome: Physical Functional Disability - Functional Capacity (METs)
Description: as for outcome 2
Time Frame: Exit at 12 weeks
Population: Exercise stress testing at exit (12 weeks) by treatment
Measure: Mean (Standard Deviation); unit: metabolism equivalents
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 14 | 13
metabolism equivalents | 6.1 (2.4) | 5.4 (2.5)
Statistical Analysis 1: Comparison: Hormone Replacement Therapy vs Placebo; Test type: Superiority or Other; p = 0.49, Wilcoxon rank sum test

11. Secondary Outcome: Physical Functional Disability - Functional Capacity (Metabolism Equivalents)
Description: Physical functional disability measured by exercise stress testing. Functional capacity was measured as metabolism equivalents (METs), exercise duration, and exercise-induced chest pain.
Time Frame: Baseline
Population: Exercise stress testing at baseline by treatment
Measure: Mean (Standard Deviation); unit: metabolism equivalents
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 17 | 16
metabolism equivalents | 6.1 (3.0) | 5.8 (2.1)
Statistical Analysis 1: Comparison: Hormone Replacement Therapy vs Placebo; Test type: Superiority or Other; p = 0.77, Wilcoxon rank sum test

12. Secondary Outcome: Physical Functional Disability - Functional Capacity (Metabolism Equivalents)
Description: as for outcome 11
Time Frame: Exit (12 weeks)
Population: Exercise stress testing at exit (12 weeks) by treatment
Measure: Mean (Standard Deviation); unit: metabolism equivalents
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 14 | 13
metabolism equivalents | 6.1 (2.4) | 5.4 (2.5)
Statistical Analysis 1: Comparison: Hormone Replacement Therapy vs Placebo; Test type: Superiority or Other; p = 0.40, Wilcoxon rank sum test

13. Secondary Outcome: Physical Functional Disability - Functional Capacity (Exercise Induced ST Segment Depression)
Description: Physical functional disability measured by exercise stress testing. Functional capacity was measured as metabolism equivalents (METs), exercise duration, and exercise-induced chest pain.
  In electrocardiography, the ST segment connects the QRS complex and the T wave and has duration of 80 to 120 ms. It should be essentially level with the PR and TP segment. The normal ST segment has a slight upward concavity. Flat, downsloping, or depressed ST segment may indicate coronary ishcemia. Positive treadmill exercise stress test (>1.0 mm horizontal / downsloping or >1.5 upsloping ST segment depression measured 0.08 msec after the J point).
Time Frame: Baseline
Population: Exercise stress testing at baseline by treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 17 | 16
mm | -0.79 (0.78) | -0.79 (0.47)
Statistical Analysis 1: Comparison: Hormone Replacement Therapy vs Placebo; Test type: Superiority or Other; p = 0.99, Wilcoxon rank sum test

14. Secondary Outcome: Physical Functional Disability - Functional Capacity (Stress Induced ST Segment Depression)
Description: as for outcome 13
Time Frame: Exit (12 weeks)
Population: Exercise stress testing at exit (12 weeks) by treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 14 | 13
mm | -1.05 (0.98) | -0.63 (0.29)
Statistical Analysis 1: Comparison: Hormone Replacement Therapy vs Placebo; Test type: Superiority or Other; p = 0.21, Wilcoxon rank sum test

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Hormone Replacement Therapy | Placebo
Serious Adverse Events (participants affected / at risk) | 2/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hormone Replacement Therapy (N=18) | Placebo (N=19)
Hospitalization for angina and a stroke (Cardiac disorders) | 1 (1) | 0 (0) — Hospitalization for angina an a stroke
Hospitalizaton for biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) — Hospitalizaton for biliary colic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No